CLINICAL TRIAL: NCT02038738
Title: 68Ga-DOTATATE PET Scan Imaging in Patients With Neuroendocrine Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Richard J. Campeau, M.D., FACNM, Professor of Radiology and Internal Medicine, Ochsner Health System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 68Ga-DOTATATE
Record Dates: First submitted 2014-01-14; First posted 2014-01-17 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Neuroendocrine; Neuroendocrine Tumor; Neuroendocrine Cancer; Neuroendocrine Carcinoma; Carcinoid; Carcinoid Tumor; Islet Cell Tumor; Apudoma
Keywords: gallium; Ga; PET Scan
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoma, Neuroendocrine; Carcinoid Tumor; Adenoma, Islet Cell; Apudoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Scan (Experimental): We will perform 68Ga-DOTATATE PET scans on subjects.
  Interventions: Drug: 68Ga-DOTATATE will be given in tracer doses and injected intravenously to image tumors by Positron Emission Tomography.

INTERVENTIONS:
Drug: 68Ga-DOTATATE will be given in tracer doses and injected intravenously to image tumors by Positron Emission Tomography.

SUMMARY:
Neuroendocrine cancer is an unusual disease and often goes undetected by routine imaging. The 68Ga-DOTATATE PET Scan is a novel scanning method that may have improved sensitivity and resolution specifically for neuroendocrine tumors. Patients with neuroendocrine tumors will be imaged with this agent and it will be compared to conventional imaging methods to determine the safety and efficacy of this radiopharmaceutical.

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of neuroendocrine tumor or suspected SSTR positive tumors by 111In-Octreotide scan, 18FDG-PET, or MRI of the abdomen where clinically indicated
* At least 18 years of age
* Able to provide informed consent
* Karnofsky performance score greater than 50
* Females of childbearing potential must have a negative pregnancy test at screening/baseline

Exclusion Criteria:

* Serum creatinine > 2.0 mg/dL
* Hepatic enzyme levels more than 3 times upper limit of normal
* Known severe allergy or hypersensitivity to IV radiographic contrast
* Use of any other investigational product or device within 30 days prior to dosing, or known requirement for any other investigational agent prior to completion of all scheduled study assessments
* Patients with a body weight of 400 pounds or more or not able to enter the bore of the PET/CT scanner due to BMI, because of the compromise in image quality with CT, PET/CT, and MRI that will result
* Inability to lie still for the entire imaging time (e.g. cough, severe arthritis, etc.)
* Inability to complete the needed investigational standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Recognized concurrent active infection
* Previous systemic or radiation treatment for another cancer of any type within the last 2 years
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2014-03; Primary Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 5 years

SECONDARY OUTCOMES:
Number of lesions detected by 68Ga-DOTATATE compared to conventional imaging techniques | 5 years
We want to determine if the 68Ga-DOTATATE PET Scan changes care plans compared to conventional imaging/diagnostic techniques (Octreoscan, MRI, CT) | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Medical Center - Kenner, Kenner, Louisiana, United States